CLINICAL TRIAL: NCT00916591
Title: Effect of Prokinetic Drugs During the Administration of Enteral Nutrition
Brief Title: Prokinetic Drugs and Enteral Nutrition
Acronym: prokinetics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Van De Winkel Nele MD, UZBrussels
Other Study IDs: UZBrussels; 2009-012342-23
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Critically Ill; Enteral Nutrition
Keywords: gastroesophageal reflux; respiratory aspiration
MeSH Terms: conditions — Critical Illness; Gastroesophageal Reflux; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to compare the effect of two drugs that can help in the prevention of regurgitation during the administration of enteral nutrition and define which one is the most effective.

DETAILED DESCRIPTION:
Two prokinetic drugs (metoclopramide and erythromycin) will be compared during the administration of enteral nutrition in critically ill patients. We would like to know which one is the most effective in preventing regurgitation and risk of aspiration, which is a common complication of enteral nutritional support. This will be evaluated by measuring gastric residue every six hours.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients
* intubated
* mechanically ventilated
* 18 or older age
* enterally fed

Exclusion Criteria:

* prokinetic drugs before start study
* allergy to study medication
* interactions odf study medication with other drugs
* recent gastro-intestinal surgery
* history of esophagectomy or gastrectomy
* suspicion of gastrointestinal perforation
* myasthenia gravis
* liver dysfunction
* less than 7 days in study
* gastro- or jejunostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients, intubated and mechanically ventilated, 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-09

CONTACTS AND LOCATIONS:
Locations (1):
- UZBrussels, Jette, Belgium